CLINICAL TRIAL: NCT03088553
Title: Etude Observationnelle Comparant l'efficacité du GANciclovir en Fonction de l'EXposition Sanguine au médicament
Brief Title: Observational Study Comparing the Efficacy of Ganciclovir as a Function of Blood Exposure to the Drug During a Curative or Preemptive Treatment
Acronym: GANEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_9773
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Solid Organ Transplantation
Keywords: Ganciclovir; trough concentrations; CMV viral load; safety; Solid organ transplantation (heart, kidney or liver)
MeSH Terms: conditions — Multiple Acyl Coenzyme A Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

INTERVENTIONS:
Drug: Therapeutic Drug Monitoring — Trough concentration of ganciclovir and viral load measurement at each follow-up visit.

SUMMARY:
This study aims to better define the target range of ganciclovir trough concentrations by investigating the relationship between ganciclovir concentration and the time to undetectable CMV-DNA load, in preemptive and curative treatments by (val)ganciclovir.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether higher concentrations of ganciclovir can reduce the time of negation of the CMV-DNA load.

Secondary objectives are to determine the concentration-toxicity relationship of ganciclovir and the relationship between concentrations of ganciclovir and apparition of CMV gene mutations responsible of drug resistance.

Each week, trough concentrations of ganciclovir are measured, associated with control of CMV-DNA load and all biological analysis currently necessary for the monitoring of the infection.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years-old
* Solid organ transplanted patients needing a treatment by oral or intravenous (val)ganciclovir
* Non-opposition to participate in the study.

Exclusion Criteria:

* pregnancy
* opposition to participate in the study
* incapable person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ transplanted patients with CMV reactivation or CMV disease.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2024-06-21 (Estimated)

PRIMARY OUTCOMES:
Time to CMV viral load negativity as a function of the median of trough concentrations of ganciclovir | through study completion, an average of 1 year
  Duration of patient follow-up for the CMV infection

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France